CLINICAL TRIAL: NCT01751308
Title: A Phase 1-2 Dose Finding, Safety and Efficacy Study of Cabazitaxel in Pediatric Patients With Refractory Solid Tumors Including Tumors of the Central Nervous System
Brief Title: Safety and Efficacy of Cabazitaxel in Pediatric Patients With Refractory Solid Tumors Including Central Nervous System Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED12689; U1111-1128-5704 (Other: UTN)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-06

CONDITIONS: Malignant Solid Tumor - Malignant Nervous System Neoplasm
MeSH Terms: interventions — cabazitaxel; XRP6258

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Phase 1: Cabazitaxel 20 mg/m^2 (Experimental): Cabazitaxel 20 mg/m^2 intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression (DP) or discontinuation due to adverse event (AE) or death (from any cause).
  Interventions: Drug: Cabazitaxel (XRP6258)
- Phase 1: Cabazitaxel 25 mg/m^2 (Experimental): Cabazitaxel 25 mg/m^2 IV infusion on Day 1 of each 21-day cycle until DP or discontinuation due to AE or death (from any cause).
  Interventions: Drug: Cabazitaxel (XRP6258)
- Phase 1: Cabazitaxel 30 mg/m^2 (Experimental): Cabazitaxel 30 mg/m^2 IV infusion on Day 1 of each 21-day cycle until DP or discontinuation due to AE or death (from any cause).
  Interventions: Drug: Cabazitaxel (XRP6258)
- Phase 1: Cabazitaxel 35 mg/m^2 (Experimental): Cabazitaxel 35 mg/m^2 IV infusion on Day 1 of each 21-day cycle until DP or discontinuation due to AE or death (from any cause).
  Interventions: Drug: Cabazitaxel (XRP6258)
- Phase 2: Cabazitaxel 30 mg/m^2 (Experimental): Cabazitaxel at the maximum tolerated dose (MTD) as determined in phase 1 (30 mg/m^2) IV infusion on Day 1 of each 21-day cycle until DP or discontinuation due to AE or death (from any cause).
  Interventions: Drug: Cabazitaxel (XRP6258)

INTERVENTIONS:
Drug: Cabazitaxel (XRP6258) — Pharmaceutical form: Injection Route of administration: Intravenous
  Other Names: Jevtana

SUMMARY:
Primary Objectives:

Phase 1 Part:

To determine the dose limiting toxicity (DLT) and the maximum tolerated dose (MTD) of cabazitaxel as a single agent in pediatric participants with recurrent or refractory solid tumors including tumors of the central nervous system.

Phase 2 Part:

To determine the objective response rate (complete and partial response) and the duration of response to cabazitaxel as a single agent in participants with recurrent or refractory high grade glioma (HGG) or diffuse intrinsic pontine glioma (DIPG).

Secondary Objectives:

Phase 1 Part:

To characterize the safety and tolerability of cabazitaxel in participants with recurrent or refractory solid tumors including tumors of the central nervous system.

To characterize the pharmacokinetic (PK) profile of cabazitaxel in participants with recurrent or refractory solid tumors including tumors of the central nervous system.

To evaluate preliminary anti-tumor activity that may be associated with cabazitaxel in participants with recurrent or refractory solid tumors including tumors of the central nervous system.

Phase 2 Part:

To characterize the safety and tolerability of cabazitaxel in participants with recurrent or refractory HGG or DIPG.

To estimate progression free survival in participants with recurrent or refractory HGG or DIPG.

To estimate overall survival in participants with recurrent or refractory HGG or DIPG.

To characterize the plasma PK profile of cabazitaxel in participants with recurrent or refractory HGG or DIPG.

DETAILED DESCRIPTION:
The study duration will include a period for inclusion of up to 3 weeks and a 3-week treatment cycle(s). The participants may continue treatment until disease progression, unacceptable toxicity or willingness to stop followed by a minimum of 30-day follow-up.

ELIGIBILITY:
Inclusion criteria:

Phase 1 Part (dose escalation): Participants with a histologically confirmed solid tumor including tumors of the central nervous system that was recurrent or refractory and for which no further effective standard treatment was available. All participants must had measurable disease. Participants with diffuse pontine glioma were eligible without a biopsy after evidence of progressive disease post radiation therapy.

Phase 2 Part (safety and activity): Participants with recurrent or refractory high grade glioma or diffuse intrinsic pontine glioma for whom no further effective therapy was available. All participants must had measurable disease. Participants with diffuse pontine glioma were eligible without a biopsy after evidence of progressive disease post radiation therapy. Participants with a grade III or grade IV glioma must had pathologic confirmation either at the time of initial diagnosis or at the time of recurrence.

Participants aged ≥2 years and ≤18 years

Participants met the body surface area (BSA) requirements to be eligible:

1. Minimal BSA requirements for a particular dose level;
2. During the Phase 1 part participants must had a BSA <2.1 m² at the time of enrollment
3. During the Phase 2 part participants with a BSA ≥2.1 m² were eligible, however the actual dose of cabazitaxel for these participants were adjusted to a maximum dose calculated with (capped at) the BSA of 2.1 m²

Performance status by:

1. Lansky score ≥60 (participants ≤10 years of age)
2. Karnofsky score ≥60% (participants >10 years of age) Participants who were unable to walk because of paralysis, but who were mobile in a wheelchair, were considered ambulatory for the purpose of assessing the performance score.

Participants must had adequate liver, renal and marrow function as defined below:

1. Total bilirubin ≤1.0 x the upper limit of normal (ULN) for age
2. AST (SGOT) and ALT (SGPT) ≤2.5 x ULN
3. Serum creatinine ≤1.5 x ULN for age or creatinine clearance ≥60 mL/min/1.73 m²
4. Absolute neutrophil count ≥1.0x10^9 /L
5. Platelets ≥75x10^9/L (transfusion independent)
6. Hemoglobin ≥8.0 g/dL (could be transfused)

Female participants of child-bearing potential must had a negative pregnancy test ≤7 days before starting cabazitaxel treatment.

Male and female participants of reproductive potential must agreed to use adequate contraception prior to study entry, for the duration of study participation and for 6 months following the last dose of cabazitaxel.

Written informed consent/assent prior to any study-specific procedures. Consent must be obtained from the participant and/or parent(s) or legal guardian(s) and the signature of at least one parent or guardian was required. Investigators also obtained assent of participants according to local, regional or national guidelines.

Participants must have recovered from the acute toxic effects of all prior therapy to ≤ grade 1 before entering the study.

Exclusion criteria:

Prior treatment within the following timeframes:

1. Systemic anti-cancer treatment within 3 weeks (6 weeks for nitrosourea, mitomycin and monoclonal antibodies including bevacizumab)
2. Surgery or smaller field radiation therapy within 4 weeks
3. Treatment with an investigational agent within 4 weeks or within 5 half-lives of the agent, whichever was longer Craniospinal or other large field radiation therapy (defined as >25% of bone marrow irradiated) within 6 months prior to the first dose.

Prior systemic radioisotope therapy (this did not include diagnostic imaging or radioimmunoconjugates lacking myelosuppressive properties) or total body irradiation.

Prior bone marrow or stem cell transplant

Participants with any clinically significant illness that, in the investigator's opinion, could not be adequately controlled with appropriate therapy, would compromise a participant's ability to tolerate cabazitaxel or result in inability to assess toxicity. This included, but was not limited to uncontrolled intercurrent illness including ongoing or active infection, cardiac disease, renal impairment, planned surgery or psychiatric illness/social situations that would limit compliance with study requirements.

Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency-syndrome (AIDS)-related disease Known history of hepatitis C or known active hepatitis B infection. Pregnant or breast feeding women Treatment with strong inhibitors or strong inducers of CYP3A4 or enzyme inducing anti-epileptic drugs (EIAED) within 14 days prior to first dose of cabazitaxel and for the duration of study. Non-EIAEDs were permitted.

Known history of hypersensitivity to taxanes or polysorbate 80 or G-CSF. Participation in another interventional clinical trial and/or concurrent treatment with any investigational drug.

Participants not able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2013-02; Primary Completion 2015-07 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- United States (12):
  - Investigational Site Number 840009, Phoenix, Arizona
  - Investigational Site Number 840013, Los Angeles, California
  - Investigational Site Number 840014, Palo Alto, California
  - Investigational Site Number 840007, Aurora, Colorado
  - Investigational Site Number 840011, Washington D.C., District of Columbia
  - Investigational Site Number 840005, Orlando, Florida
  - Investigational Site Number 840012, Chicago, Illinois
  - Investigational Site Number 840010, Baltimore, Maryland
  - Investigational Site Number 840002, Boston, Massachusetts
  - Investigational Site Number 840003, New York, New York
  - Investigational Site Number 840006, Houston, Texas
  - Investigational Site Number 840008, Seattle, Washington
- Investigational Site Number 124001, Toronto, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 12 centers between February 2013 and March 2015.
Pre-assignment Details: Phase I was a dose escalation part of Cabazitaxel to determine maximum tolerated dose (MTD). Phase 2 was efficacy and safety evaluation of Cabazitaxel at the MTD, determined in Phase 1.
Groups:
- Phase 1: Cabazitaxel 20 mg/m^2: Cabazitaxel 20 mg/m^2 intravenous (IV) infusion on Day 1 of each 21-day cycle until disease progression (DP) or discontinuation due to adverse events (AE) or death (from any cause).
- Phase 2: Cabazitaxel 30 mg/m^2: Cabazitaxel at the MTD as determined in phase 1 (30 mg/m^2) IV infusion on Day 1 of each 21-day cycle until DP or discontinuation due to AE or death (from any cause).
Period: Phase 1
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 | Phase 1: Cabazitaxel 25 mg/m^2 | Phase 1: Cabazitaxel 30 mg/m^2 | Phase 1: Cabazitaxel 35 mg/m^2 | Phase 2: Cabazitaxel 30 mg/m^2
Started | 6 | 3 | 7 | 7 | 0 (Phase 1 and Phase 2 were separate populations.)
Completed | 6 (DP, AE and death were considered as completed (defined in protocol)) | 3 (DP, AE and death were considered as completed (defined in protocol)) | 7 (DP, AE and death were considered as completed (defined in protocol)) | 7 (DP, AE and death were considered as completed (defined in protocol)) | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 | Phase 1: Cabazitaxel 25 mg/m^2 | Phase 1: Cabazitaxel 30 mg/m^2 | Phase 1: Cabazitaxel 35 mg/m^2 | Phase 2: Cabazitaxel 30 mg/m^2
Started | 0 | 0 | 0 | 0 | 16 (Phase 1 and Phase 2 were separate populations.)
Completed | 0 | 0 | 0 | 0 | 16 (DP, AE and death were considered as completed (defined in protocol))
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated (AT)/safety population was defined as all registered participants who actually received at least 1 dose or part of a dose of the investigational medicinal product (IMP).
Groups:
- Phase 1: Cabazitaxel 20 mg/m^2: Cabazitaxel 20 mg/m^2 IV infusion on Day 1 of each 21-day cycle until DP or discontinuation due to AE or death (from any cause).
- Total: Total of all reporting groups
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 | Phase 1: Cabazitaxel 25 mg/m^2 | Phase 1: Cabazitaxel 30 mg/m^2 | Phase 1: Cabazitaxel 35 mg/m^2 | Phase 2: Cabazitaxel 30 mg/m^2 | Total
Number analyzed (Participants) | 6 | 3 | 7 | 7 | 16 | 39
Age, Customized [Number; unit: participants]
  2-4 years | 0 | 0 | 2 | 0 | 2 | 4
  5-6 years | 2 | 1 | 0 | 1 | 4 | 8
  7-11 years | 1 | 1 | 3 | 5 | 4 | 14
  12-18 years | 3 | 1 | 2 | 1 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 1 | 2 | 8 | 16
  Male | 1 | 3 | 6 | 5 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose of Cabazitaxel
Description: MTD was highest dose level of cabazitaxel at which no more than 1 of 6 evaluable participants experienced dose limiting toxicities (DLT). DLT defined as an AE or abnormal laboratory values related to study treatment: hematologic DLTs: any Grade(G)4 hematologic toxicity except neutropenia G4 lasting≤7 days,G3 or 4 febrile neutropenia except G3 or 4 febrile neutropenia in absence of granulocyte-colony stimulating factor prophylaxis, G4 thrombocytopenia; non-hematologic DLTs:any G≥3 non-hematologic toxicity except G3 nausea or G3 or4 vomiting, G3 or4 diarrhea,G3 or4 dehydration,G3 fatigue lasting≤7 days, inadequately treated hypersensitivity reactions, elevated transaminases<10* upper limit of normal of ≤7 days, re-treatment delay of>2 weeks due to delayed recovery from toxicity related to study treatment to baseline G or≤ G1(except for alopecia) and platelet transfusion during Cycle1. Grades based on National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Cycle 1 (21 days)
Population: DLT evaluable population defined as a subset of participants in the Phase 1 part of the study from the AT population who received the first dose of cabazitaxel and had sufficient safety evaluations or experienced a DLT during Cycle 1.
Measure: Number; unit: mg/m^2
Groups:
- Phase 1: Overall Population: Cabazitaxel 20 mg/m^2, 25 mg/m^2, 30 mg/m^2 or 35 mg/m^2 IV infusion on Day 1 of each 21-day cycle until DP or discontinuation due to AE or death (from any cause).
Arm/Group | Phase 1: Overall Population
Number analyzed (Participants) | 23
mg/m^2 | 30

2. Primary Outcome: Phase 2: Percentage of Participants With Objective Response (OR)
Description: OR in participants was defined as the participants with a Complete Response (CR) or Partial Response (PR) after 3 cycles of cabazitaxel treatment and maintained for at least 4 weeks. CR and PR were based on modified response assessment in neuro-oncology (RANO) criteria for participants with CNS tumors. CR was defined as disappearance of all target lesions. PR was defined as ≥50% decrease in the sum of the products of the two perpendicular diameters of target lesions, compared to the baseline measurement.
Time Frame: Baseline, every 9 weeks until DP or death due to any cause (maximum duration: 12.1 weeks)
Population: Efficacy evaluable population was subset of AT population with measurable disease with a baseline and at least one post-baseline tumor evaluation.Number of participants analyzed=participants with available data for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Cabazitaxel 30 mg/m^2
Number analyzed (Participants) | 11
percentage of participants
  CR | 0
  PR | 0

3. Primary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR defined as time (in days) from date of first response until date of first documented progressive disease (PD) or death (from any cause), whichever came first. If progression or death was not observed, participant was censored at the date of participant's last progression-free tumor assessment prior to study cut-off date. PD as per RANO criteria was defined as ≥ 25% increase in the product of perpendicular diameters of any target lesion, taking as reference the smallest product observed since the start of treatment or the appearance of one or more new lesions, or worsening neurologic status not explained by causes unrelated to tumor progression (example, anticonvulsant or corticosteroid toxicity, electrolyte disturbances, sepsis, hyperglycemia, presumed post-therapy swelling etc.) plus any increase in tumor cross-sectional area (or tumor volume).
Time Frame: Baseline, every 9 weeks until DP or death due to any cause (maximum duration: 12.1 weeks)
Population: Due to no objective responses in Stage 1 of Phase 2, the analysis of duration of response was not performed.Hence, the data is not reported.
Arm/Group | Phase 2: Cabazitaxel 30 mg/m^2
Number analyzed (Participants) | 0

4. Secondary Outcome: Phase 1 and 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had a causal relationship with the treatment. Treatment emergent adverse events (TEAEs) were defined as AEs that developed or worsened in grade or became serious during the on-treatment period which was defined as the period from the time of first dose of cabazitaxel until 30 days following the last administration of cabazitaxel.
Time Frame: Baseline up to DP or death due to any cause (maximum duration: 112.1 weeks for Phase 1 and 12.1 weeks for Phase 2)
Population: Analysis was performed on safety population (AT population).
Measure: Number; unit: participants
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 | Phase 1: Cabazitaxel 25 mg/m^2 | Phase 1: Cabazitaxel 30 mg/m^2 | Phase 1: Cabazitaxel 35 mg/m^2 | Phase 2: Cabazitaxel 30 mg/m^2
Number analyzed (Participants) | 6 | 3 | 7 | 7 | 16
participants | 6 | 3 | 7 | 7 | 16

5. Secondary Outcome: Phase 1: Number of Participants With Objective Response
Description: OR in participants was defined as the participants with a CR or PR after 3 cycles of cabazitaxel treatment and maintained for at least 4 weeks as assessed by response evaluation criteria in solid tumors (RECIST) version 1.1 and RANO criteria for CNS tumors. For solid tumors, as per RECIST 1.1, CR defined as disappearance of all target and non-target lesions (any pathological lymph nodes, must had reduction in short axis to <10 mm); PR defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. For CNS tumors, as per RANO criteria, CR defined as disappearance of all target and non-target lesions; PR defined as a ≥50% decrease in the sum of the products of the two perpendicular diameters of target lesions, compared to baseline measurement.
Time Frame: Baseline, every 9 weeks until DP or death due to any cause (maximum duration: 112.1 weeks)
Population: Analysis was performed on efficacy evaluable population. Number of participants analyzed=participants with available data for this endpoint.
Measure: Number; unit: participants
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 | Phase 1: Cabazitaxel 25 mg/m^2 | Phase 1: Cabazitaxel 30 mg/m^2 | Phase 1: Cabazitaxel 35 mg/m^2
Number analyzed (Participants) | 5 | 3 | 7 | 7
participants | 1 | 0 | 0 | 0

6. Secondary Outcome: Phase 1 and 2: Pharmacokinetics (PK) Parameter of Cabazitaxel: Area Under the Plasma Concentration (AUC) Versus Time Curve
Description: Blood samples for PK parameters were collected at 5 minutes before end of infusion (EOI), 10 minutes, 30 minutes, 3 hours, 7 hours and 71 hours after the EOI on Day 1 of Cycle 1.
Time Frame: Day 1 of Cycle 1: 5 minutes before EOI up to 71 hours after the EOI
Population: PK population (for both Phase 1 and Phase 2 parts of the study) included all participants who received treatment on Day 1 of Cycle 1 and had at least one post-dose PK sample. Number of participants analyzed=participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Groups:
- Phase 1 and 2: Cabazitaxel 30 mg/m^2: Cabazitaxel 30 mg/m^2 IV infusion on Day 1 of each 21-day cycle (at the MTD dose determined in Phase 1) in Phase 1 and Phase 2 until DP or discontinuation due to AE or death (from any cause).
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 | Phase 1: Cabazitaxel 25 mg/m^2 | Phase 1 and 2: Cabazitaxel 30 mg/m^2 | Phase 1: Cabazitaxel 35 mg/m^2
Number analyzed (Participants) | 6 | 3 | 20 | 2
ng.h/mL | 669.5 (430.6) | 879.0 (414.7) | 876.7 (359.9) | 1002.5 (277.9)

7. Secondary Outcome: Phase 1 and 2: PK Parameter of Cabazitaxel: Total Plasma Clearance (CL)
Description: Blood samples for PK parameters were collected at 5 minutes before EOI, 10 minutes, 30 minutes, 3 hours, 7 hours and 71 hours after the EOI on Day 1 of Cycle 1.
Time Frame: Day 1 of Cycle 1: 5 minutes before EOI up to 71 hours after the EOI
Population: Analysis was performed on PK population (for both Phase 1 and Phase 2 parts of the study). Number of participants analyzed=participants with available data for this endpoint.
Measure: Mean (Standard Deviation); unit: L/h/m^2
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 | Phase 1: Cabazitaxel 25 mg/m^2 | Phase 1 and 2: Cabazitaxel 30 mg/m^2 | Phase 1: Cabazitaxel 35 mg/m^2
Number analyzed (Participants) | 6 | 3 | 20 | 2
L/h/m^2 | 36.05 (12.91) | 32.76 (12.72) | 38.70 (12.98) | 36.61 (9.98)

8. Secondary Outcome: Phase 1 and 2: PK Parameter of Cabazitaxel: Volume of Distribution at Steady State (Vss)
Description: as for outcome 7
Time Frame: Day 1 of Cycle 1: 5 minutes before EOI up to 71 hours after the EOI
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L/m^2
Groups:
- Phase 1: Cabazitaxel 25 mg/m^2: Cabazitaxel 25 mg/m^2 IV infusion on Day 1 of each 21-day cycle until DP or discontinuation due to AEor death (from any cause).
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 | Phase 1: Cabazitaxel 25 mg/m^2 | Phase 1 and 2: Cabazitaxel 30 mg/m^2 | Phase 1: Cabazitaxel 35 mg/m^2
Number analyzed (Participants) | 6 | 3 | 20 | 2
L/m^2 | 3391.72 (686.79) | 3301.96 (351.55) | 3371.30 (975.98) | 1488.75 (1179.11)

9. Secondary Outcome: Phase 1 and 2: PK Parameter of Cabazitaxel: Maximum Plasma Concentration Observed (Cmax)
Description: as for outcome 7
Time Frame: Day 1 of Cycle 1: 5 minutes before EOI up to 71 hours after the EOI
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 | Phase 1: Cabazitaxel 25 mg/m^2 | Phase 1 and 2: Cabazitaxel 30 mg/m^2 | Phase 1: Cabazitaxel 35 mg/m^2
Number analyzed (Participants) | 6 | 3 | 20 | 2
ng/mL | 204.864 (189.864) | 283.657 (242.970) | 256.734 (127.931) | 233.290 (0.127)

10. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: The PFS was defined as the time (in months) from the date of first dose administration until the date of first documented PD or death (from any cause), whichever came first. If progression or death was not observed, the participant was censored at the date of the participant's last progression-free tumor assessment prior to the study cut-off date. PD as per RANO criteria was defined as ≥25% increase in the product of perpendicular diameters of any target lesion, taking as reference the smallest product observed since the start of treatment or the appearance of one or more new lesions, or worsening neurologic status not explained by causes unrelated to tumor progression (example, anticonvulsant or corticosteroid toxicity, electrolyte disturbances, sepsis, hyperglycemia, presumed post-therapy swelling etc) plus any increase in tumor cross-sectional area (or tumor volume). The analysis was performed by Kaplan-Meier method.
Time Frame: Baseline, every 9 weeks until DP or death due to any cause (maximum duration: 12.1 weeks)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Cabazitaxel 30 mg/m^2
Number analyzed (Participants) | 11
months | 1.3 [0.6 to 2.1]

11. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of first dose administration until the date of death (from any cause). If death was not observed, the participant was censored at the earliest of the last date the participant was known to be alive and the study cut-off date. The analysis was performed by Kaplan-Meier method.
Time Frame: Baseline up to death or study cut-off (maximum duration: 12.1 weeks)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Cabazitaxel 30 mg/m^2
Number analyzed (Participants) | 11
months | 2.7 [1.7 to 4.5]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (112.1 weeks for Phase 1 and 12.1 weeks for Phase 2) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during 'on treatment period' (time from first dose of study drug to last dose of study drug + 30 days). Analysis was performed on safety population.
Arm/Group | Phase 1: Cabazitaxel 20 mg/m^2 | Phase 1: Cabazitaxel 25 mg/m^2 | Phase 1: Cabazitaxel 30 mg/m^2 | Phase 1: Cabazitaxel 35 mg/m^2 | Phase 2: Cabazitaxel 30 mg/m^2
Serious Adverse Events (participants affected / at risk) | 4/6 | 1/3 | 5/7 | 3/7 | 12/16
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 7/7 | 7/7 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Cabazitaxel 20 mg/m^2 (N=6) | Phase 1: Cabazitaxel 25 mg/m^2 (N=3) | Phase 1: Cabazitaxel 30 mg/m^2 (N=7) | Phase 1: Cabazitaxel 35 mg/m^2 (N=7) | Phase 2: Cabazitaxel 30 mg/m^2 (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Death (General disorders) | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 0 | 0 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 3
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Stoma site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Brain herniation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Nerve root compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Cabazitaxel 20 mg/m^2 (N=6) | Phase 1: Cabazitaxel 25 mg/m^2 (N=3) | Phase 1: Cabazitaxel 30 mg/m^2 (N=7) | Phase 1: Cabazitaxel 35 mg/m^2 (N=7) | Phase 2: Cabazitaxel 30 mg/m^2 (N=16)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 1 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eyelid pain (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4 | 1 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 2 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3 | 2 | 4
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Device occlusion (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 2 | 3 | 3
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 2
Rectal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Candida test positive (Investigations) | 0 | 0 | 1 | 0 | 0
Coronavirus test positive (Investigations) | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 2 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Accessory nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 2 | 2
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebellar ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Cerebellar syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Cranial nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 3
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 1 | 1 | 2 | 4
Hemiparesis (Nervous system disorders) | 2 | 1 | 0 | 0 | 3
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypoglossal nerve disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
VIIIth nerve lesion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
VIth nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Deja vu (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.